CLINICAL TRIAL: NCT04845412
Title: Hearing Screening Outcomes of Two Screening Tests in Newborns of Gestational Diabetic and Non-diabetic Mothers: a Prospective, Controlled Study
Brief Title: Hearing Screening Outcomes of Two Screening Tests in Newborns of Gestational Diabetic Mothers
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Esra Gulen Yıldız, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: CGDMP2020
Record Dates: First submitted 2021-04-10; First posted 2021-04-15 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Gestational Diabetes; Hearing Loss
Keywords: Gestational diabetes; Hearing loss; Newborns
MeSH Terms: conditions — Diabetes, Gestational; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children of GDM parents: Children of mothers who have gestational diabetes mellitus
  Interventions: Diagnostic Test: Hearing screening tests
- Children of non-diabetic parents: Children of mothers without diabetes
  Interventions: Diagnostic Test: Hearing screening tests

INTERVENTIONS:
Diagnostic Test: Hearing screening tests — Our study was conducted in accordance with the National Hearing Screening Test Protocol. The newborns had transient evoked otoacoustic emissions (TEOAE) with "click" stimulus as a hearing screening test in the first three days after birth, using Otometrics Madsen Accuscreen S/N: 36484 (USA) device.

SUMMARY:
In this study, the investigators have aimed to investigate whether GDM is a risk factor for hearing impairment in newborns. To the investigators knowledge, this study is the first prospective, controlled study on this subject.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is an increasingly frequent condition in the world causing significant morbidity and mortality. GDM is a metabolic disease that develops in pregnancy, and may result in complications in the pregnant women, similar to other patients with diabetes. The prevalence of GDM varies in relation with the population and the diagnostic criteria. Diabetes affects 6-9% of pregnant women; 99% of the cases have GDM, and diabetes is diagnosed before pregnancy in the remaining 1% [(pre-gestational diabetes mellitus (pre-GDM)]. Hearing loss is one of the most common birth defect in newborns. The incidence of congenital hearing impairment is 2-3 per 1000 births. Early diagnosis and treatment is very important for the development of auditory pathways and protection of cognitive functions. Therefore, newborn hearing screening programs have been in use in a number of countries. Transient evoked otoacoustic emissions (TEOAE) and auditory brainstem response (ABR) have been identified as basic convenient and applicable tools for neonatal screening of hearing.

Suboptimal glycemic control during pregnancy has adverse fetal effects. Congenital malformations, preterm birth and neonatal respiratory distress in the newborn are more common, at varying rates, pre-GDM and GDM. Compared to the normal population, the risk of congenital malformations is 1.9-10 fold higher in presence of pre-GDM, and 1.1-1.3 fold higher in presence of GDM. Despite our awareness on these important complications, the effect of intrauterine hyperglycemia on hearing of the newborn has not yet been studied in detail. Diabetes mellitus (DM) often causes hearing impairment, however little is known whether GDM is an antenatal risk factor for cochlear damage and hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Women with gestational diabetes
* Women without diabetic pregnancy

Exclusion Criteria:

* Admitted to the neonatal intensive care unit for more than five days
* Perinatal asphyxia
* Craniofacial abnormalities
* İntrauterine infections
* Hyperbilirubinemia requiring exchange transfusion
* Very low birth weight (<1500 g)
* Gestational hypertension
* Preeclampsia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with gestational diabetes Women without diabetic pregnancy
Study Population: Women with gestational diabetes and women without diabetic pregnancy
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of Hearing loss | One year
  Rate of newborns who failed hearing screening tests

CONTACTS AND LOCATIONS:
Overall Officials: Esra Gulen Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No